CLINICAL TRIAL: NCT00153998
Title: Open, Randomized, Multicenter, Randomized Phase II Trial Comparing the Combination of Cetuximab With Oxaliplatin/5-FU/FA Versus the Combination of Cetuximab With Irinotecan/5-FU/FA as Neoadjuvant Treatment in Patients With Non-Resectable Colorectal Liver Metastases
Brief Title: Cetuximab in Neoadjuvant Treatment of Non-Resectable Colorectal Liver Metastases (CELIM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. Claus-Henning Köhne, now: Klinikum Oldenburg gGmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELIM
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2007-04

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Cetuximab; Oxaliplatin; Irinotecan; 5-FU; Chemotherapy; Resection; Liver resection; Neoadjuvant
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Hepatectomy; Irinotecan; Fluorouracil; Leucovorin; Folfox protocol; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cetuximab and FOLFIRI
  Interventions: Drug: Cetuximab; Procedure: Liver resection; Drug: Cetuximab and FOLFIRI
- 2 (Active Comparator): Cetuximab and FOLFOX
  Interventions: Drug: Cetuximab; Procedure: Liver resection; Drug: Cetuximab and FOLFOX

INTERVENTIONS:
Drug: Cetuximab
Procedure: Liver resection
Drug: Cetuximab and FOLFIRI — Cetuximab 400 mg/m² (2.0 h i.v.) (first dose only), followed by:
  Cetuximab 250 mg/m² (1.0 h i.v.) weekly
  Irinotecan 180 mg/m² (2.0 h i.v.) all compounds day 1, repeated at day 15 Folinic acid (D,L) 400 mg/m² (2.0 h i.v.) 5-FU 400 mg/m² (bolus i.v.) 5-FU 2400 (-3000) mg/m² (46 h i.v.)
  Other Names: Cetuximab(C225, Erbitux®, Merck KGaA); Irinotecan (irinotecan HCl, CPT-11 or Campto®, Aventis); 5-Fluorouracil (5-FU); Folinic acid (FA, i.e. Leucovorin®, Wyeth)
  Arms: 1
Drug: Cetuximab and FOLFOX — Cetuximab 400 mg/m² (2.0 h i.v.) (first dose only), followed by:
  Cetuximab 250 mg/m² (1.0 h i.v.) weekly
  Oxaliplatin 100 mg/m² (2.0 h i.v.) all compounds day 1, repeated at day 15 Folinic acid (D,L) 400 mg/m² (2.0 h i.v.) 5-FU 400 mg/m² (bolus i.v.) 5-FU 2400 (-3000) mg/m² (46 h i.v.)
  Other Names: Cetuximab(C225, Erbitux®, Merck KGaA); Oxaliplatin (L-OHP, Eloxatin®, Sanofi-Synthelabo); 5-Fluorouracil (5-FU); Folinic acid (FA, i.e. Leucovorin®, Wyeth)
  Arms: 2

SUMMARY:
General Objectives:

* To test the feasibility of neoadjuvant treatment with cetuximab/chemotherapy followed by liver resection
* To determine the optimal combination (cetuximab/FOLFOX versus cetuximab/FOLFIRI) for further trials in preoperative chemotherapy

DETAILED DESCRIPTION:
Patients with liver metastasis will be screened for this study. Eligible patients will complete the pretreatment evaluation including an abdominal CT scan that will be presented to the local surgeon and the radiologist for proving of resectability of hepatic lesions. Additionally, CT scans will be reviewed by three reference surgeons. In case of non-resectability, as defined above, CT- or ultrasound- guided biopsy of one of the liver metastases will be performed, unless biopsy material is available from prior biopsy of one of the liver metastases.

Instead of an ultrasound-guided biopsy, a CT-guided biopsy may be performed.

Formalin-fixed, paraffin embedded metastatic tissue will be sent to reference laboratory (Prof. Störkel, Wuppertal) for immunohistochemical analysis of EGFR- expression.

Additionally tissue will be stored in "RNA later" for gene expression analysis if agreed by the patient.

Additionally, the primary tumor will be collected and sent to the reference laboratory for analysis of EGFR- expression (if agreement of the patient exists).

Patients will be randomized to a combination of:

Cetuximab/FOLFIRI (irinotecan/5-FU/FA) or Cetuximab/FOLFOX6 (oxaliplatin/5-FU/FA)

All patients receive a four month treatment (eight cycles) of the allocated treatment.

Resection is planned after completion of neoadjuvant treatment and should be performed between 4 and 6 weeks after the last dose of chemotherapy. Probes of the resected material (in liquid nitrogen and paraffin embedded material will be collected).

If a resection is not possible after eight administrations of chemotherapy, chemotherapy will be continued until tumor progression (maximal duration of treatment 2 years) and the patient will be evaluated for a potential resection every two months.

After resection, postoperative treatment is planned for 3 months (6 cycles). Treatment start is planned between 4 and 8 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-resectable, histologically confirmed, synchronous or metachronous colorectal liver metastases. Patients with non-resectable metastases are defined as; patients with five or more liver metastases; and/or patients with liver metastases that are technically non-resectable (local surgeon in cooperation with local radiologist will define non-resectability on the basis of remaining functional liver tissue, infiltration of all liver veins, infiltration of both liver arteries, both portal branches or both bile ducts).
* Patients with simultaneous liver metastases are eligible, if the primary tumor has been resected at least 1 month prior to chemotherapy.
* Karnofsky Performance Status ≥ 80
* Informed consent
* Adequate bone marrow function, liver and renal function (neutrophils > 1.5 x 10^9/l; thrombocytes > 100 x 10^9/l; hemoglobin > 8.0 g/l; bilirubin ≤ 1.5 x upper limit of normal [ULN] and not increasing more than 25% within the last 4 weeks; ALAT and ASAT < 5 x UNL; serum creatinine ≤ 1.5 x UNL)
* Age ≥ 18 years

Exclusion Criteria:

* Any evidence of extrahepatic metastases, lymph node metastases and primary tumor recurrence
* Prior chemotherapy (except adjuvant chemotherapy with an interval of ≥ 6 months)
* Previous exposure to EGFR (epidermal growth factor receptor)-targeting therapy
* Radiotherapy or major abdominal or thoracic surgery (excluding diagnostic biopsy or port implantation) ≤ 4 weeks before study entry
* Concurrent systemic immune therapy, chemotherapy, or hormone therapy
* Investigational agents or participation in clinical trials within 30 days before start of the treatment in study
* Clinically relevant coronary disease or myocardial infarction within 12 months before study entry
* Peripheral neuropathy > CTC grade I
* Inflammatory bowel disease
* Previous malignancy (except colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
* History of severe psychiatric illness
* Drug or alcohol abuse
* Breast feeding or pregnant women, no effective contraception if risk of conception exists (male and female patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Tumor response, defined as partial and complete response according to RECIST (Response Evaluation Criteria in Solid Tumors) - criteria in the intention-to-treat [ITT-] population

SECONDARY OUTCOMES:
Rate of R0 liver resection (ITT- population)
Progression free survival (ITT- population)
Disease free survival after resection (ITT- population)
Overall survival (ITT- population)
Safety (all patients that received any study drug)
Molecular predictive markers for response and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Claus-Henning Köhne, Prof. Dr., Principal Investigator — Klinikum Oldenburg GmbH, Dr.-Eden-Str.10; 26133 Oldenburg; Gunnar Folprecht, Dr., Principal Investigator — University Hospital Dresden, Fetscherstr. 74, 01307 Dresden, Germany
Locations (21):
- Medizinische Universitaet Wien, Universitaetsklinik für Chirurgie, Vienna, Austria
- Germany (20):
  - Kreiskrankenhaus Aschersleben, Aschersleben
  - Charite-Campus Benjamin Franklin, Innere Medizin, Berlin
  - Charite-Campus, Virchow-Klinikum, Innere Medizin, Berlin
  - Allgemeines Krankenhaus Celle, Celle
  - University Hospital "Carl Gustav Carus", Dresden
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Universitaet Erlangen-Nuernberg, Chirurgie, Erlangen
  - Westdeutsches Tumorzentrum, Universitaetsklinikum Essen, Essen
  - Johann Wolfgang Goethe Universitaet, Chirurgie, Frankfurt am Main
  - Westpfalz-Klinikum GmbH Innere Medizin I, Kaiserslautern
  - UKSH Campus Kiel, II. Medizinische Klinik, Kiel
  - Staedtisches Klinikum Magdeburg-Olvenstedt, Magdeburg
  - Universitaetsklinik Mannheim gGmbH, III. Medizinische Klinik, Mannheim
  - Klinikum Grosshadern, III. Medizinische Klinik, München
  - Klinikum Oldenburg GmbH, Oldenburg
  - Klinikum Passau, II. Medizinische Klinik, Passau
  - Klinikum der Hansestadt Stralsund GmbH, Medizinische Klinik, Stralsund
  - Krankenhaus der Barmherzigen Brueder Trier, Chirurgie, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Chirurgie, Würzburg

REFERENCES:
- [Derived] Folprecht G, Gruenberger T, Bechstein W, Raab HR, Weitz J, Lordick F, Hartmann JT, Stoehlmacher-Williams J, Lang H, Trarbach T, Liersch T, Ockert D, Jaeger D, Steger U, Suedhoff T, Rentsch A, Kohne CH. Survival of patients with initially unresectable colorectal liver metastases treated with FOLFOX/cetuximab or FOLFIRI/cetuximab in a multidisciplinary concept (CELIM study). Ann Oncol. 2014 May;25(5):1018-25. doi: 10.1093/annonc/mdu088. Epub 2014 Feb 27. PMID 24585720
- [Derived] Folprecht G, Gruenberger T, Bechstein WO, Raab HR, Lordick F, Hartmann JT, Lang H, Frilling A, Stoehlmacher J, Weitz J, Konopke R, Stroszczynski C, Liersch T, Ockert D, Herrmann T, Goekkurt E, Parisi F, Kohne CH. Tumour response and secondary resectability of colorectal liver metastases following neoadjuvant chemotherapy with cetuximab: the CELIM randomised phase 2 trial. Lancet Oncol. 2010 Jan;11(1):38-47. doi: 10.1016/S1470-2045(09)70330-4. Epub 2009 Nov 26. PMID 19942479